CLINICAL TRIAL: NCT01633450
Title: Bioavailability of Zinc From Rice Biofortified With 70Zn and Rice Extrinsically Labeled With 70Zn in Young Adults: a Randomized, Single-blind Study
Brief Title: Zinc Absorption From Biofortified Rice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: HNL/CTC12-Reis
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
MeSH Terms: interventions — Zinc

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Zinc biofortified rice (Experimental)
  Interventions: Other: Zinc biofortified rice
- Rice extrinsically fortified with zinc (Active Comparator)
  Interventions: Other: Rice extrinsically fortified with zinc

INTERVENTIONS:
Other: Zinc biofortified rice — 1.12 mg zinc per meal
  Arms: Zinc biofortified rice
Other: Rice extrinsically fortified with zinc — 1.12 mg zinc per meal
  Arms: Rice extrinsically fortified with zinc

SUMMARY:
One of the newest strategies to combat micronutrient deficiencies is the biofortification of staple foods, where higher levels of minerals are obtained through breeding of staple crops. The aim of this study is to evaluate zinc absorption from a rice biofortified with zinc when compared with a control rice fortified with zinc just before consumption.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of 18 to 45 years old
* Body Mass Index in the range of 19 to 25
* No mineral and vitamin supplements two weeks prior to the study and during the whole duration of the study

Exclusion Criteria:

* Any metabolic, gastrointestinal or chronic disease (according to the subjects own statement)
* Long-term medication during the whole study (except for contraceptives)
* Pregnancy
* Lactation
* Intention to become pregnant during the course of the study
* Lack of safe contraception
* Consumption of mineral and vitamin supplements within 2 weeks prior to 1st - Earlier participation in any nutrition study using Zn stable isotopes as well as participation in any other clinical study within the last 30 days and during this study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Fractional absorption of zinc | 33 days
  Fractional absorption of zinc is estimated by using the double isotope tracer ratio technique by administering 67Zn as oral and 70Zn as intravenous stable isotopes.The urinary enrichment with both isotopes is measured in a spot urine sample by inductively coupled plasma mass spectrometry.

CONTACTS AND LOCATIONS:
Locations (1):
- ETH Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Brnic M, Wegmuller R, Melse-Boonstra A, Stomph T, Zeder C, Tay FM, Hurrell RF. Zinc Absorption by Adults Is Similar from Intrinsically Labeled Zinc-Biofortified Rice and from Rice Fortified with Labeled Zinc Sulfate. J Nutr. 2016 Jan;146(1):76-80. doi: 10.3945/jn.115.213421. Epub 2015 Dec 16. PMID 26674764